CLINICAL TRIAL: NCT03167125
Title: Participatory Research to Advance Colon Cancer Prevention
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other); AltaMed Health Services Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 1U01MD010665-01 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; cancer screening; pragmatic trial; boot camp translation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I: The investigators will conduct a three-arm patient-randomized trial to compare 1) usual care, 2) automated prompts, and 3) automated plus live prompts. (Number of Arms: 3)
  Phase II: This spread trial will use a stepped-wedge design, which is a variant of a crossover randomized trial, where clinics cross over from usual practice to the best practices program. In the stepped-wedge design, a baseline period controls for the level and rate of change of the outcomes prior to program implementation and the staggered implementation minimizes confounding due to changes in the secular trend. By randomizing practices to when they receive an intervention instead of whether they receive it, the stepped wedge design ensures that all practices eventually receive the intervention, an important consideration for clinic leadership. Furthermore, the wedge-defined clusters act as their own controls as they each receive both intervention conditions. (Number of Arms: 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated Prompts (Active Comparator): Patients randomized to this arm will receive automated prompts to complete and return the FIT kit.
  Interventions: Other: Automated Prompts
- Automated Plus Live Prompts (Active Comparator): Patients randomized to this arm will receive automated prompts plus linguistically and culturally tailored live prompts to complete and return the FIT kit.
  Interventions: Other: Automated Plus Live Prompts
- Usual Care (No Intervention): Patients randomized to this arm will receive usual care screening opportunities per recommended colorectal cancer screening guidelines.

INTERVENTIONS:
Other: Automated Prompts — This intervention is an automated data-driven program, using automated phone calls, text messages, and/or emails, for delivering FIT kit prompts to patients due for colorectal cancer screening. The specific components of the intervention are forthcoming and will be determined using a community-based participatory research approach known as boot camp translation which seeks input from patients and providers.
  Arms: Automated Prompts
Other: Automated Plus Live Prompts — This intervention is a higher-intensity program, using automated data-driven prompts plus linguistically and culturally tailored live prompts, for delivering FIT kit messages to patients due for colorectal cancer screening. The specific components of the intervention are forthcoming and will be determined using a community-based participatory research approach known as boot camp translation which seeks input from patients and providers.
  Arms: Automated Plus Live Prompts

SUMMARY:
The overall goal of this study is to test strategies to raise rates of colorectal cancer screening among the Latino population in a federally qualified health center that operates multiple clinics. This intervention study will test automated and live prompts to a direct-mail fecal testing program in two phases.

In Phase I (Years 01 - 02), the investigators will tailor and define intervention components using a community-based participatory research approach called boot camp translation (BCT). The ultimate design of the intervention will be defined by patient and provider feedback from BCT. The investigators will then conduct a three-arm patient-randomized comparative effectiveness trial in two pilot clinics to compare 1) automated prompts (i.e., automated phone calls, text messages) to alert and remind patients to complete screening, 2) live prompts (i.e., live phone calls), and 3) a combination approach of automated plus live prompts.

In Phase II (Years 03 - 05), the investigators will spread and test the spread of the adapted intervention to additional clinics within the partnering health center using a two-arm main trial.

Both phases will be guided by an advisory group of clinicians, researchers, policy makers, and patients.

DETAILED DESCRIPTION:
The study will fulfill the following aims:

Aim 1: Develop personalized messages (e.g., phone scripts, text messages, patient portal prompts) and define an intervention using boot camp translation to increase colon cancer screening among Latino populations.

Aim 2: Assess the reach, effectiveness, and differences by subgroup (e.g., preferred language) of a three-arm colorectal cancer screening program among Latino FQHC patients, in 2 clinics, through a patient randomized-controlled trial.

In addition to Usual Care, the arms are:

* Automated Prompts-an automated data-driven program for delivering FIT kit prompts (using automated phone calls, text messages, and/or emails) to patients due for colorectal cancer screening.
* Automated Plus Live Prompts-a higher-intensity program using automated, data-driven strategies for delivering FIT kit prompts plus linguistically and culturally tailored live prompts.

Aim 3: Test the spread of the program across additional clinics using a two-arm randomized approach and develop an implementation guide that includes outreach materials, strategies for incorporating patient input, and resources.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 50-75 years and not up-to-date with colorectal cancer screening

Exclusion Criteria:

* Persons having colorectal disease (e.g., ulcerative colitis or colectomy), personal history of colorectal cancer or colorectal disease, end-stage or life threatening diseases or, those known to be under hospice care or living in a skilled nursing facility may be excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27580 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Increased colorectal cancer screening rates | Up to 4 years (study period)
  Fecal testing completion

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Coronado, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- AltaMed Health Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coronado GD, Nyongesa DB, Escaron AL, Petrik AF, Thompson JH, Smith D, Davis MM, Schneider JL, Rivelli JS, Laguna T, Leo MC. Effectiveness and Cost of an Enhanced Mailed Fecal Test Outreach Colorectal Cancer Screening Program: Findings from the PROMPT Stepped-Wedge Trial. Cancer Epidemiol Biomarkers Prev. 2023 Nov 1;32(11):1608-1616. doi: 10.1158/1055-9965.EPI-23-0597. PMID 37566431
- [Derived] Schneider JL, Rivelli JS, Vaughn KA, Thompson JH, Petrik AF, Escaron AL, Coronado GD. Implementing an enhanced mailed FIT program to improve CRC screening at a federally qualified health center: experiences of patients and staff. Transl Behav Med. 2023 Sep 28;13(10):757-767. doi: 10.1093/tbm/ibad025. PMID 37210075
- [Derived] Davis MM, Schneider JL, Petrik AF, Miech EJ, Younger B, Escaron AL, Rivelli JS, Thompson JH, Nyongesa D, Coronado GD. Clinic Factors Associated With Mailed Fecal Immunochemical Test (FIT) Completion: The Difference-Making Role of Support Staff. Ann Fam Med. 2022 Mar-Apr;20(2):123-129. doi: 10.1370/afm.2772. PMID 35346927
- [Derived] Coronado GD, Nyongesa DB, Petrik AF, Thompson JH, Escaron AL, Younger B, Harbison S, Leo MC. Randomized Controlled Trial of Advance Notification Phone Calls vs Text Messages Prior to Mailed Fecal Test Outreach. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2353-2360.e2. doi: 10.1016/j.cgh.2020.07.053. Epub 2020 Jul 30. PMID 32739569
- [Derived] Coronado GD, Thompson JH, Petrik AF, Nyongesa DB, Leo MC, Castillo M, Younger B, Escaron A, Chen A. Patient-Refined Messaging for a Mailed Colorectal Cancer Screening Program: Findings from the PROMPT Study. J Am Board Fam Med. 2019 May-Jun;32(3):318-328. doi: 10.3122/jabfm.2019.03.180275. PMID 31068396
- [Derived] Thompson JH, Davis MM, Leo MC, Schneider JL, Smith DH, Petrik AF, Castillo M, Younger B, Coronado GD. Participatory Research to Advance Colon Cancer Prevention (PROMPT): Study protocol for a pragmatic trial. Contemp Clin Trials. 2018 Apr;67:11-15. doi: 10.1016/j.cct.2018.02.001. Epub 2018 Feb 9. PMID 29408304